CLINICAL TRIAL: NCT06677528
Title: Gender-specific Evaluation of Symptom Awareness in Female Versus Male Patients with Severe Aortic Stenosis
Acronym: AWARE
Status: Active, not recruiting | Type: Observational
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Other Study IDs: HDZ-KA_022_TR
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-09

CONDITIONS: Aortic Stenosis; Female; Male
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients undergoing TAVR or SAVR
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire on Aortic Valve Disease, HADS-D, SCL-27, MLHFQ

SUMMARY:
The objectives of this single center cross-sectional cohort study are to compare symptoms and disease perception of male and female patients with severe aortic stenosis.

DETAILED DESCRIPTION:
Background Aortic valve stenosis is a common valvular disease that increases with age and is associated with a poor prognosis when severe (1-3). Treatment options include surgical or interventional replacement of the aortic valve . Awareness of aortic valve stenosis in the general population is low (2% in Europe) (4). Auscultation as a simple screening tool is relatively underused. This leads to a clear underdiagnosis of aortic stenosis especially in patients with only minor or no complaints. In addition, several studies show a marked gender discrepancy: women tend to be diagnosed later, checked less regularly for asymptomatic vitium, and operated on or intervened later (5-7). One possible reason for this could be gender-specific symptom perception. For example, women perceive pain more variably, sensitively, and intensely than men and report more painful conditions. Related to a possible myocardial infarction, women show a greater number of additional, ostensibly nonbreast-related pain symptoms regardless of the presence of chest pain. Both female patients and practitioners are less likely to attribute their prodromal symptoms to heart disease compared with men. Women are generally at higher risk for affective disorders (e.g., depression, anxiety disorders) than men, with greater susceptibility varying with age (8-10).

Literature

1. Andell P, Li X, Martinsson A, Andersson C, Stagmo M, Zoller B, et al. Epidemiology of valvular heart disease in a Swedish nationwide hospital-based register study. Heart 2017;103:1696-1703. https://doi.org/10.1136/heartjnl-2016-310894
2. Marciniak A, Glover K, Sharma R. Cohort profile: prevalence of valvular heart disease in community patients with suspected heart failure in UK. BMJ Open 2017;7:e012240. https://doi.org/10.1136/bmjopen-2016-012240
3. Nkomo VT, Gardin JM, Skelton TN, Gottdiener JS, Scott CG, Enriquez-Sarano M. Burden of valvular heart disease: a population-based study. Lancet 2006;368: 1005-1011. https://doi.org/10.1016/S0140-6736(06)69208-8.
4. Gaede L, Di Bartolomeo R, van der Kley F, Elsasser A, Iung B, Mollmann H. Aortic valve stenosis: what do people know? A heart valve disease awareness survey of over 8,800 people aged 60 or over. EuroIntervention 2016;12:883-889. https://doi.org/10.4244/ EIJY16M06_02.
5. Vassileva CM, McNeely C, Mishkel G, Boley T, Markwell S, Hazelrigg S. Gender differences in long-term survival of Medicare beneficiaries undergoing mitral valve operations. Ann Thorac Surg 2013;96:1367-1373. https://doi.org/10.1016/j.athoracsur. 2013.04.055 62.
6. Tanguturi VK, Bhambhani V, Picard MH, Armstrong K, Wasfy JH. Echocardiographic surveillance of valvular heart disease in different sociodemographic groups. JACC Cardiovasc Imaging 2019;12:751-752. https://doi.org/10.1016/j.jcmg.2018.05.025
7. Tastet L, Kwiecinski J, Pibarot P, Capoulade R, Everett RJ, Newby DE, et al. Sex-related differences in the extent of myocardial fibrosis in patients with aortic valve stenosis. JACC Cardiovasc Imaging 2020;13:699-711. https://doi.org/10.1016/j.jcmg.2019.06.014
8. Pieretti S, Di Giannuario A, Di Giovannandrea R, Marzoli F, Piccaro G, Minosi P, Aloisi AM. Gender differences in pain and its relief. Ann Ist Super Sanita. 2016 Apr-Jun;52(2):184-9. doi: 10.4415/ANN_16_02_09. PMID: 27364392.
9. Lichtman JH, Leifheit EC, Safdar B, Bao H, Krumholz HM, Lorenze NP, Daneshvar M, Spertus JA, D'Onofrio G. Sex Differences in the Presentation and Perception of Symptoms Among Young Patients With Myocardial Infarction: Evidence from the VIRGO Study (Variation in Recovery: Role of Gender on Outcomes of Young AMI Patients). Circulation. 2018 Feb 20;137(8):781-790. doi: 10.1161/CIRCULATIONAHA.117.031650. PMID: 29459463; PMCID: PMC5822747.
10. Faravelli C, Alessandra Scarpato M, Castellini G, Lo Sauro C. Gender differences in depression and anxiety: the role of age. Psychiatry Res. 2013 Dec 30;210(3):1301-3. doi: 10.1016/j.psychres.2013.09.027. epub 2013 Oct 2. PMID: 24135551.

ELIGIBILITY:
Inclusion Criteria:

* • Indication for surgical or interventional aortic valve replacement for aortic stenosis as consented by the local heart team

  * Age> 18 years
  * Patient is willing and able to complete the surveys in German language

Exclusion Criteria:

* • Additional procedures such as coronary bypass surgery, any surgery on another than the aortic valve, aortic surgery

  * PCI performed within the last 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About n=800 Patients who are admitted for surgical or interventional replacement of aortic stenosis complete the following questionnaires:
  1. HADS - D
  2. SCL - 27
  3. MLHFQ
  4. Demographic data
  5. AWARE - Symptoms of aortic stenosis
Sampling Method: Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-07-31 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Questionnaires completed | From enrollment to the end of FU at 4 weeks

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Clinic for General and Interventional Cardiology/Angiology, Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Clinic for Thoracic and Cardiovascular Surgery, Herz- und Diabeteszentrum NRW, Bad Oeynhausen

IPD SHARING:
Plan to Share IPD: No